CLINICAL TRIAL: NCT07316439
Title: Clinical Outcomes of ER-Positive to Negative Conversion Versus Triple-Negative Breast Cancer (TNBC): Evidence From a 18F-fluoroestradiol Positron Emission Tomography/Computed Tomography (18F-FES PET/CT) Guided Propensity-Score-Matched Study
Brief Title: Comparison Between ER Loss and Triple-Negative Breast Cancer Guided by 18F-FES PET/CT in Metastatic Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-36
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ER negative conversion group: 82 patients with functional ER loss detected by FES-PET at metastatic sites before first-line treatment
- mTNBC: A total of 115 contemporaneous patients with metastatic TNBC at initial diagnosis

SUMMARY:
This study aimed to compare survival outcomes and clinical characteristics between ER loss and metastatic triple-negative breast cancer (mTNBC) patients, exploring the prognostic implications of dynamic ER changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer (according to International Classification of Diseases 10th Revision) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
* MBC patients who underwent 18F-FES PET/CT at the Fudan University Shanghai Cancer Center between 2017 and 2023
* Patients diagnosed with primary ER-positive tumor and who were yet to receive any systemic therapy during the advanced stage
* Contemporaneous patients with metastatic TNBC at initial diagnosis

Exclusion Criteria:

* Patients with incomplete medical records and those diagnosed with secondary primary tumors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MBC patients with ER-positive primary tumor who detected negative ER expression in metastatic disease using 18F-FES PET/CT at Fudan University Shanghai Cancer Center. Contemporaneous patients with metastatic TNBC at initial diagnosis at Fudan University Shanghai Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 6 weeks

SECONDARY OUTCOMES:
Overall Response Rate | 6 weeks
Disease Control Rate | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided